CLINICAL TRIAL: NCT04239482
Title: Longer-term Effects of a Novel Nutritional Combination on Muscle Insulin Sensitivity and Mitochondrial Function, and Vascular Function in Abdominally Obese Subjects
Brief Title: Nutritional Supplementation and Insulin Sensitivity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to covid-19 pandemic
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: METC 19-085
Record Dates: First submitted 2019-12-20; First posted 2020-01-27 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2020-09

CONDITIONS: Nitric Oxide; Insulin Sensitivity; Vascular Function; L-arginine; Nitrate / Nitrite
MeSH Terms: conditions — Insulin Resistance | interventions — Arginine; Nitrates; Nitrites

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-arginine + Nitrate/Nitrite (Experimental): Subjects will receive 1 L-arginine tablet per day and drink 35 mL of beetroot juice for 8 weeks.
  Interventions: Dietary Supplement: L-arginine + Nitrate / Nitrite
- Placebo (Placebo Comparator): Subjects will receive 1 cellulose tablet per day and drink 35 mL of nitrate/nitrite depleted beetroot juice for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-arginine + Nitrate / Nitrite — Longer-term supplementation (8 weeks)
  Arms: L-arginine + Nitrate/Nitrite
Dietary Supplement: Placebo — Longer-term supplementation (8 weeks)
  Arms: Placebo

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a progressive disease and early intervention and prevention strategies are therefore very important. An important early hallmark in the development of T2DM is insulin resistance. Since the majority of postprandial glucose disposal occurs in skeletal muscle, improving muscle insulin sensitivity will thus have a major impact on disease prevention. Abdominally obese men and women have an increased risk to develop T2DM, and are also characterized by an impaired vascular function. This may hamper proper delivery of insulin, glucose and oxygen to muscles, thereby contributing to - and possibly causing - muscle insulin resistance. Earlier it has been shown that supplementation with L- arginine improves vascular function by improving nitric oxide (NO) bioavailability. These NO- mediated beneficial effects on vascular function may improve delivery of insulin, glucose and oxygen to the muscle tissue, thereby improving muscle insulin sensitivity and mitochondrial function. However, the doses needed of this amino acid cannot be provided by regular diets or supplements, also due to the bitter taste of L-arginine. Alternatively, smaller amounts of L- arginine with a specific combination of other nutritional components (i.e. nitrate and nitrite), which are already part of the regular diet and support alternative pathways to improve NO- mediated vascular function, may also induce beneficial effects. The investigators now hypothesize that in abdominally obese adults with impaired fasting glucose concentrations L-arginine combined with nitrate/nitrite increases muscle insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 50-70 years
* Men and postmenopausal (two or more years after last menstruation) women
* Waist circumference for men 3 102 cm and for women 3 88 cm (abdominally obese)
* Impaired fasting glucose concentrations (between 5.6 - 7.0 mmol/L in accordance with the American Diabetes Association guidelines for prediabetes) at two screening visits
* Fasting serum total cholesterol < 8.0 mmol/L
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit
* Willingness to give up the use of antibacterial mouth wash or antibacterial toothpaste, chewing-gum and tongue-scraping during the study

Exclusion Criteria:

* Current smoker, or smoking cessation < 12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* More than 3 alcoholic consumptions per day
* Use of dietary supplements known to interfere with the main study outcomes as judged by the principal investigators
* Use of anticoagulant drugs or drugs to treat blood pressure, lipid/glucose metabolism
* Use of an investigational product within another biomedical intervention trial within the previous 1-month
* Intolerance or allergy to the ingredients of the intervention products
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease (COPD), inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity | Change between 8-week placebo and 8-week intervention period
  Muscle insulin sensitivity

SECONDARY OUTCOMES:
Change in muscle metabolism | Change between 8-week placebo and 8-week intervention period
  Mitochondrial activity in muscle tissue
Change in physical functioning (1) | Change between 8-week placebo and 8-week intervention period
  6 meter walking test
Change in physical functioning (2) | Change between 8-week placebo and 8-week intervention period
  Timed up and go test
Change in physical functioning (3) | Change between 8-week placebo and 8-week intervention period
  Handgrip strength test
Change in physical functioning (4) | Change between 8-week placebo and 8-week intervention period
  Isokinetic muscle strength (BIODEX measurement)
Change in vascular function (1) | Change between 8-week placebo and 8-week intervention period
  Flow-mediated vasodilation of the brachial artery
Change in vascular function (2) | Change between 8-week placebo and 8-week intervention period
  Pulse wave analysis
Change in vascular function (3) | Change between 8-week placebo and 8-week intervention period
  Pulse wave velocity
Change in vascular function (4) | Change between 8-week placebo and 8-week intervention period
  Retinal microvascular calibers (Artery-to-Vein ratio)
Change in cardiometabolic risk markers (1) | Change between 8-week placebo and 8-week intervention period
  Plasma markers for low-grade systemic inflammation (CRP)
Change in cardiometabolic risk markers (2) | Change between 8-week placebo and 8-week intervention period
  Plasma markers for endothelial dysfunction (NOx)
Change in cardiometabolic risk markers (3) | Change between 8-week placebo and 8-week intervention period
  24-h Systolic and Diastolic blood pressure
Change in continuous insulin sensitivity | Change between 8-week placebo and 8-week intervention period
  36-h plasma glucose values

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Joris, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No